CLINICAL TRIAL: NCT01842373
Title: A Double-Blind, Randomized, Split-Face Comparison Trial on Topical Anesthetic Agents Prior to Fractional Skin Resurfacing
Brief Title: Comparison Study on Topical Anesthetic Agents (LMX4 and BLT) Prior to Fractional Skin Resurfacing
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding not secured
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Solta Medical (Industry)
Responsible Party: Principal Investigator, Charlene Lam, Resident Physician, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 41491
Record Dates: First submitted 2013-04-25; First posted 2013-04-29 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Pain
Keywords: topical anesthetics; laser resurfacing
MeSH Terms: conditions — Pain | interventions — Receptors, Leukotriene B4; Benzocaine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LMX4 (Experimental): 3 g of LMX4 will be applied to one half of the face for 60 minutes
  Interventions: Drug: BLT
- BLT (Active Comparator): 3 g of BLT will be applied to half of face for 60 minutes
  Interventions: Drug: LMX4

INTERVENTIONS:
Drug: LMX4
  Other Names: LMX 4 (Lidocaine 4%)
  Arms: BLT
Drug: BLT
  Other Names: BLT (Benzocaine 20%, lidocaine 6%, tetracaine 4%)
  Arms: LMX4

SUMMARY:
The purpose of this research study is to test which topical anesthesia: LMX4 (Lidocaine 4%) or BLT (Benzocaine 20%, Lidocaine 6%, and Tetracaine 4%) is more effective in reducing discomfort during treatment with the Fraxel DUAL 1550/1927 (Solta Medical, Hayward, CA). No studies have been done on the effectiveness of LMX4 versus BLT using the Fraxel DUAL, although individually LMX4, BLT, and the Fraxel DUAL have been studied extensively.

The hypothesis is that there will be no clinical difference between the two topical anesthetics.

DETAILED DESCRIPTION:
Lasers can be effectively utilized for facial rejuvenation, reduction of photoinduced rhytides, and dyschromia. Topical anesthetics are used to minimize the discomfort associated with laser induced thermal pain. There are currently several formulations of topical anesthesia. However, studies comparing the products are limited especially for the new formulations that claim increased efficacy and faster onset.

LMX4 (Ferndale Laboratories, Ferndale, Michigan) is over the counter topical anesthesia. It is 4% lidocaine that has been formulated into multilamellar vesicles containing several lipid bilayers. This unique liposomal-based delivery system has been reported to deliver a greater concentration of drug. This results in a longer duration of activity and faster onset of action without requiring occlusion.4 Liposomes assist with drug penetration because the skin is lipid bilayer that can encapsulate the drug.

BLT is a compounded topical anesthetic containing 20% benzocaine, 6% lidocaine, and 4% tetracaine. It is commonly prescribed as topical anesthesia. All BLT products will be compounded at the University Physicians Center Pharmacy to ensure safety and uniformity. Anecdotally, some physicians claim it is the topical anesthesia of choice prior to laser surgery.

The objective of the study is to evaluate the clinical efficacy of topical anesthetic compounds prior to fractional skin resurfacing.

ELIGIBILITY:
Inclusion Criteria:

* At least 28 subjects will be included in this study.
* Subjects capable of giving informed consent.
* Patients 18 years of age and older will be included in this study.
* Any patient seeking Fraxel DUAL1550/1927 (Solta Medical) treatment on the face for rhytids, photoaging, hyperpigmentation, and acne scarring at the Hershey Medical Center dermatology clinics will be asked to participate.

Exclusion Criteria:

* Age <18
* Allergy to lidocaine or tetracaine
* Women who are pregnant or breast-feeding
* Patients with cardiac or respiratory disease, seizure disorders, or neuropathy
* Patients currently taking anxiolytics and opiates

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2013-09 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Patient Assessment of Pain | Immediately after laser treatment
  A pain assessment will be performed on both halves of the face by utilizing a standard 10 cm visual analog pain scale (VAS).

CONTACTS AND LOCATIONS:
Locations (1):
- Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States